CLINICAL TRIAL: NCT04869345
Title: Feasibility of a Positive Affect Skills Intervention for Reducing Racial Disparities in Pain Management
Brief Title: Positive Affect as a Source of Resilience for Adults in Chronic Pain
Acronym: LARKSPUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Cornell University (Other); Wake Forest University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-06022291; 5P30AG022845 (NIH); 5U24AG058556 (NIH)
Record Dates: First submitted 2021-04-10; First posted 2021-05-03 (Actual); Results first posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Geriatric; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LARKSPUR intervention (Experimental): Lessons in Affect Regulation to Keep Stress and Pain UndeR control
  Interventions: Behavioral: LARKSPUR
- Attention Control Condition (No Intervention): Daily emotion reporting/no intervention

INTERVENTIONS:
Behavioral: LARKSPUR — This intervention used in our prior research consists of skills training exercises designed to increase the frequency of positive affect. The 6 week intervention (5 weeks of content plus one week of home practice) consists of five components: (1) Positive events and gratitude; (2) mindfulness; (3) reappraisal; (4) strength and goals; and(5) acts of kindness. Participants will have up to 8 weeks to complete this intervention.
  Arms: LARKSPUR intervention

SUMMARY:
Fibromyalgia syndrome (FMS) is a chronic musculoskeletal condition characterized by widespread pain and tenderness, and often accompanied by impaired physical functioning, depressed mood, as well as deficits in positive affect (PA).Standard behavioral therapies typically focus on minimizing negative thoughts and emotions associated with pain and yield only modest treatment effects. Efforts are therefore needed to develop more effective psychological treatments for chronic pain by identifying new targets for intervention.

The objectives of this Stage I randomized pilot trial are to evaluate the feasibility, acceptability, and the impact of a previously developed online positive affect (PA) skills intervention -LARKSPUR (Lessons in Affect Regulation to Keep Stress and Pain UndeR control)-in a sample of Hispanic, non-Hispanic other, and non-Hispanic African American patients with fibromyalgia syndrome (FMS).

DETAILED DESCRIPTION:
Specific Aims:

Aim 1: To maximize relevance and acceptability of content and delivery of LARKSPUR intervention among patients with FMS, a chronic pain population with known deficits in PA. This aim will establish the feasibility (recruitment and retention) and acceptability (helpfulness, satisfaction, and impact) of the multicomponent LARKSPUR intervention in Hispanic, non-Hispanic African American and non-Hispanic other patients with FMS.

Aim 2: To conduct a randomized pilot trial to evaluate the impact of the LARKSPUR intervention in FMS pain (primary outcome), as well PA, depressive symptoms, physical functioning, and stress appraisals (secondary outcomes) and Aim 2a: explore racial/ethnic disparities.

For Aim 1, the study team will pilot LARKSPUR to examine feasibility and acceptability of the intervention framework by conducting frequency and descriptive statistics for enrollment rates, number of sessions completed, number of weeks required to complete the intervention, and Likert-scale items assessing satisfaction with the intervention and perceived helpfulness. For Aims 2, FMS patients (target N=90) will be randomized to receive the LARKSPUR content online or to complete daily emotion reports online (control). The researchers hypothesize that intervention participants will report more frequent PA, decreased depressive symptoms, enhanced physical functioning, improved stress appraisals, and reduced FMS pain (intensity and interference) immediately following the intervention (approximately 6-8 wks) and at 1-month post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Access to daily internet
* ≥ 50 years of age
* Able to read and understand English
* Physician diagnosis confirmation of FMS AND/OR Score ≥ 13 on the 6-item, self-report fibromyalgia screening tool
* Report having pain for at least the last three months

Exclusion Criteria:

* Cognitive impairment
* Current behavioral treatment for pain
* Enrolled in another pain study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Ong, PhD, Principal Investigator — Cornell University; Cary Reid, MD PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- NewYork-Presbyterian - Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Reduced, de-identified data sets containing data collected from patients, will be made available for secondary use at the National Archive of Computerized Data on Aging (NACDA), a division of ICPSR at the University of Michigan. NACDA is a repository of survey data on aging that has hundreds of social science research data sets available that are drawn from NIA-funded surveys and data collection efforts. NACDA has established protocols for contributors to reliably de-identify survey participants, regardless of whether they have been assembled as part of national random sample surveys or specialized registry data collection efforts. External users may be asked to provide study aims, variables requested, analytic plans, and targeted journals in their data use requests. They will also be asked to not attempt to re-identify participants, either by merging in administrative, census, medical, or other data, or by using a software program that might re-identify participants.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Background] Ong AD, Moskowitz JT, Wethington E, Addington EL, Sanni M, Goktas S, Sluys E, Swong S, Kim P, Reid MC. Lessons in Affect Regulation to Keep Stress and Pain UndeR control (LARKSPUR): Design of a randomized controlled trial to increase positive affect in middle-aged and older adults with fibromyalgia. Contemp Clin Trials. 2022 Sep;120:106880. doi: 10.1016/j.cct.2022.106880. Epub 2022 Aug 11. PMID 35964867
- [Derived] Ong A, Wilcox K, Reid MC, Wethington E, Cintron D, Addington E, Goktas S, Moskowitz J. Targeting Daily Positive Events to Improve Emotional and Functional Well-Being in Adults With Fibromyalgia: Insights From the LARKSPUR Randomized Controlled Trial. J Med Internet Res. 2024 Dec 10;26:e54678. doi: 10.2196/54678. PMID 39657168
- [Derived] Ong AD, Wilcox KT, Moskowitz JT, Wethington E, Addington EL, Sanni MO, Kim P, Reid MC. Feasibility, Acceptability, and Preliminary Efficacy of a Positive Affect Skills Intervention for Adults With Fibromyalgia. Innov Aging. 2023 Jul 13;7(10):igad070. doi: 10.1093/geroni/igad070. eCollection 2023. PMID 38094931
- See also: This manuscript describes the study design and anticipated analyses for this trial. — https://pubmed.ncbi.nlm.nih.gov/35964867/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 142 participants were recruited for the study and assessed for eligibility. Of those 142 participants, n = 22 did not meet eligibility requirements. Of the n = 120 eligible participants, n = 22 declined to participate, n = 2 were excluded by the investigators, and n = 1 was unable to access the online study platform; 95 participants met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | LARKSPUR Intervention | Attention Control Condition
Started | 49 | 46
Post-Intervention Week 11 | 43 | 43
1 Month Follow-Up Week 16 | 41 | 43
Completed | 41 | 43
Not Completed | 8 | 3
Not completed — Lost to Follow-up | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LARKSPUR Intervention | Attention Control Condition | Total
Number analyzed (Participants) | 49 | 46 | 95
Age, Customized [Count of Participants; unit: Participants]
  Between 50 and 59 years | 18 | 23 | 41
  Between 60 and 69 years | 22 | 19 | 41
  Between 70 and 79 years | 8 | 4 | 12
  >= 80 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 42 | 90
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 48 | 44 | 92
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 40 | 37 | 77
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 49 | 46 | 95
PROMIS Pain Intensity - Short Form 3a [Mean (Standard Deviation); unit: T-score] — Pain intensity T-scores measured by PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Intensity - Short Form 3a. This 3-item instrument assesses how much a person hurts. The first two items assess pain intensity over a 7-day recall period; the last item asks patients to rate their pain intensity "right now." Respondents report their pain on a 5-point scale: 1=Had no pain, 2=Mild, 3=Moderate, 4=Severe, 5=Very severe. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 36.3 to 81.8. Lower T-scores represent better outcomes.
  T-score | 63.31 (6.32) | 62.57 (5.77) | 62.95 (6.04)
PROMIS Pain Interference - Short Form 6b [Mean (Standard Deviation); unit: T-score] — Pain interference T-scores measured by PROMIS Pain Interference - Short Form 6b. This 6-item instrument measures self-reported impact of pain on a person's life and extent that pain may interfere with engagement with social, cognitive, emotional, physical, and recreational activities over a 7-day recall period. Respondents report pain interference on a 5-point scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, and 5=Very much. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 41.0 to 78.3. Lower T-scores represent better outcomes.
  T-score | 63.16 (5.99) | 62.72 (4.94) | 62.95 (5.48)
PROMIS Physical Functioning Short Form 10a [Mean (Standard Deviation); unit: T-score] — Physical function T-scores measured by PROMIS Physical Function Short Form 10a. This 10-item instrument assesses a patient's abilities and limitations with respect to everyday physical activities. Respondents report limitations on a 5-point scale: 5=Not at all, ..., 3=Somewhat, ..., 1=Cannot do, and abilities to perform activities on a 5-point scale: 5=Without any difficulty, ..., 3=With some difficulty, ..., 1=Unable to do. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 13.5 to 61.9. Higher T-scores represent better outcomes.
  T-score | 36.99 (6.03) | 37.24 (5.59) | 37.11 (5.79)
PROMIS Fatigue - Short Form 6a [Mean (Standard Deviation); unit: T-score] — Fatigue T-scores measured by PROMIS Fatigue Short Form 6a. This 6-item instrument assesses a patient's a patient's level of fatigue over a 7-day recall period. Respondents report fatigue on a 5-point scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 33.4 to 76.8. Lower T-scores represent better outcomes.
  T-score | 66.20 (7.09) | 63.31 (6.92) | 64.80 (7.12)
Depressive Symptoms (Center for Epidemiologic Studies Depression Scale Revised, CESD-R-10) [Mean (Standard Deviation); unit: units on a scale] — The 10-item version of the Center for Epidemiological Studies Depression Scale (CES-D) asks for participants to rate how often over the past week they experienced symptoms associated with depression on a 4-point scale: 0=Rarely or None of the time, 1=Some or Little of the time, 2=Moderately or Much of the time, 3=Most or Almost all the time. Mean scores range from 0.0 (rare depressive symptoms) to 3.0 (depressive symptoms most or almost all of the time).
  units on a scale | 1.23 (0.54) | 1.22 (0.55) | 1.22 (0.54)
Positive Affect (modified Differential Emotions Scale, mDES) [Mean (Standard Deviation); unit: units on a scale] — The modified Differential Emotions Scale (mDES) is a 20-item instrument that measures the extent to which a patient has experienced positive and negative emotions over a chosen time frame; in the version used in this study, we ask for emotions over the past 7 days. Respondents are asked to report the greatest amount of a given emotion on a five-point scale: 0=Not at all, 1=A little bit, 2=Moderately, 3=Quite a bit, 4=Extremely. Mean scores range from 0.0 (not at all experienced positive emotion) to 4.0 (extremely positive emotion).
  units on a scale | 1.68 (0.80) | 1.70 (0.80) | 1.69 (0.80)
Positive Affect (Positive and Negative Affect Scale, PANAS-GEN) [Mean (Standard Deviation); unit: units on a scale] — The 20-item self-report Positive and Negative Affect Scale (PANAS-GEN) asks participants to describe to what extent they feel different feelings and emotions on average. Respondents answer on a five-point scale: 0=Very slightly or not at all, 1=A little, 2=Moderately, 3=Quite a bit, 4=Extremely. Mean scores for the 10-item Positive Affect subscale range from 0.0 (very slightly or not at all positive affect) to 4.0 (extremely positive affect).
  units on a scale | 1.89 (0.72) | 1.92 (0.69) | 1.90 (0.70)
Stress Appraisal (Perceived Stress Scale) [Mean (Standard Deviation); unit: units on a scale] — The 10-item version of the Perceived Stress Scale (PSS) assesses the perception of stress over the previous month. Respondents report how often they have experienced perceived stress on a five-point scale: 0=Never, 1=Almost never, 2=Sometimes, 3=Fairly often, 4=Very often. PSS mean scores range from 0 (experienced no or minimal stress) to 4 (experienced very frequent stress).
  units on a scale | 1.86 (0.71) | 1.66 (0.61) | 1.77 (0.66)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment as Measured by Rates of Enrollment (Aim 1)
Description: Percent enrolled of total eligible participants.
Time Frame: At baseline
Population: 120 of 142 participants recruited for the study who met eligibility requirements.
Measure: Count of Participants; unit: Participants
Groups:
- All Recruited Participants Pre-Randomization: All participants recruited into the study screened for eligibility before randomization
Arm/Group | All Recruited Participants Pre-Randomization
Number analyzed (Participants) | 120
Participants
  Eligible Participants | 120
  Enrolled Participants | 95
  Declined to Participate | 22
  Excluded by the Investigators | 2
  Unable to Access the Online Study Platform | 1

2. Primary Outcome: Retention as Measured by Change in Enrollment
Description: Percentage enrolled at baseline that completed the post-intervention assessment.
Time Frame: At baseline; at week 11 (post-intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | LARKSPUR Intervention | Attention Control Condition
Number analyzed (Participants) | 49 | 46
Participants | 43 | 43
Statistical Analysis 1: Comparison: LARKSPUR Intervention vs Attention Control Condition; Test type: Superiority; p = .684, Boschloo Test — A priori threshold for statistical significance = 0.05; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.13 to 3.05] — Maximum likelihood estimate of the Odds Ratio comparing retention rate in LARKSPUR group to Attention Control group

3. Primary Outcome: Helpfulness, Satisfaction, and Impact as Assessed by Self-Report Participant Feedback Survey (Aim 1)
Description: The feedback survey collected two Likert-scale questions asking whether the participant recommends the intervention: (1) "Would you recommend LARKSPUR to a friend?" and (2) "Would you recommend LARKSPUR to someone else with chronic pain?". Both questions were measured on an 11-point scale, with 0=Definitely Not to 10=Definitely Yes. Higher scores indicate better outcomes for both questions. The two items were analyzed separately, not combined.
Time Frame: At week 11 (post-intervention)
Population: For the LARKSPUR intervention, n = 6 lost to follow-up at Week 11. For the Attention Control condition, n = 3 lost to follow-up at Week 11.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LARKSPUR Intervention | Attention Control Condition
Number analyzed (Participants) | 43 | 43
units on a scale
  Rating of Recommending Intervention to Friend | 8.89 (0.27) | 9.05 (0.25)
  Rating of Recommending Intervention to Those with Chronic Pain | 9.14 (0.23) | 8.59 (0.30)

4. Primary Outcome: Length of Intervention Time as Measured by Number of Weeks to Complete Intervention (Aim 1)
Description: Length of Intervention time as measured by number of weeks the participant took to complete the LARKSPUR intervention program.
Time Frame: At week 11 (post-intervention)
Population: For the LARKSPUR intervention, n = 6 lost to follow-up at Week 11. n = 3 participants did not complete all skills in the LARKSPUR intervention and are excluded from analysis. Attention Control group are not analyzed because they did not receive the LARKSPUR intervention.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | LARKSPUR Intervention
Number analyzed (Participants) | 40
weeks | 4.06 [4.01 to 4.17]

5. Secondary Outcome: Change in FMS Pain as Measured by PROMIS Pain Intensity - Short Form 3a (Aim 2)
Description: Pain intensity T-scores measured by PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Intensity - Short Form 3a. This 3-item instrument assesses how much a person hurts. The first two items assess pain intensity over a 7-day recall period; the last item asks patients to rate their pain intensity "right now." Respondents report their pain on a 5-point scale: 1=Had no pain, 2=Mild, 3=Moderate, 4=Severe, 5=Very severe. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 36.3 to 81.8. Lower T-scores represent better outcomes.
Time Frame: At baseline; at week 11 (post-intervention); at week 16 (1 month post intervention)
Population: For the LARKSPUR intervention, n = 6 lost to follow-up at Week 11, n = 2 lost to follow-up from Week 11 to Week 16. For the Attention Control, n = 3 lost to follow-up at Week 11. Intention-to-treat analyses were conducted for participants completing Baseline and Post-Intervention (n = 43 in LARKSPUR intervention, n = 43 in Attention Control Condition).
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | LARKSPUR Intervention | Attention Control Condition
Number analyzed (Participants) | 43 | 43
T-score
  Baseline | 63.64 [61.99 to 65.29] | 62.79 [61.01 to 64.57]
  Week 11 (Post-Intervention) | 61.22 [59.43 to 63.01] | 61.49 [59.69 to 63.28]
  Week 16 (1 month Post-Intervention): number analyzed (Participants) | 41 | 43
  Week 16 (1 month Post-Intervention) | 61.99 [60.16 to 63.82] | 61.55 [59.76 to 63.34]
Statistical Analysis 1: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 11 (Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PROMIS Pain Intensity scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.835, Mixed Models Analysis — The threshold for statistical significance was 0.05; P-value adjusted using the Kenward-Roger (1997) degrees of freedom method; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-2.80 to 2.27], Standard Error of Mean 1.28 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 2: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PROMIS Pain Intensity scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.732, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-2.12 to 3.00], Standard Error of Mean 1.29 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 3: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) in change from Week 11 (Post-Intervention) to Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PROMIS Pain Intensity scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.609, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = 0.71, 95% CI 2-sided [-2.05 to 3.47], Standard Error of Mean 1.38 — The estimated Mean Difference (Net) compares the change for the LARKSPUR intervention (Week 16 minus Week 11) minus the change for the Attention Control (Week 16 minus Week 11)

6. Secondary Outcome: Change in FMS Pain as Measured by PROMIS Pain Interference - Short Form 6b (Aim 2)
Description: Pain interference T-scores measured by PROMIS Pain Interference - Short Form 6b. This 6-item instrument measures self-reported impact of pain on a person's life and extent that pain may interfere with engagement with social, cognitive, emotional, physical, and recreational activities over a 7-day recall period. Respondents report pain interference on a 5-point scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, and 5=Very much. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 41.0 to 78.3. Lower T-scores represent better outcomes.
Time Frame: At baseline; at week 11 (post-intervention); at week 16 (1 month post intervention)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | LARKSPUR Intervention | Attention Control Condition
Number analyzed (Participants) | 43 | 43
T-score
  Baseline | 63.63 [62.02 to 65.25] | 62.78 [61.24 to 64.32]
  Week 11 (Post-Intervention) | 61.77 [60.26 to 63.28] | 62.60 [61.08 to 64.11]
  Week 16 (1 Month Post-Intervention): number analyzed (Participants) | 41 | 43
  Week 16 (1 Month Post-Intervention) | 62.11 [60.57 to 63.66] | 60.73 [59.22 to 62.25]
Statistical Analysis 1: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 11 (Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PROMIS Pain Interference scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.445, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-2.97 to 1.31], Standard Error of Mean 1.08 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 2: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PROMIS Pain Interference scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.209, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = 1.38, 95% CI 2-sided [-0.78 to 3.54], Standard Error of Mean 1.09 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 3: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) in change from Week 11 (Post-Intervention) to Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PROMIS Pain Interference scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.063, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = 2.21, 95% CI 2-sided [-0.12 to 4.54], Standard Error of Mean 1.17 — [estimate comment as in outcome 5, analysis 3]

7. Secondary Outcome: Change in Physical Functioning as Measured by PROMIS Physical Functioning Short Form 10a (Aim 2)
Description: Physical function T-scores measured by PROMIS Physical Function Short Form 10a. This 10-item instrument assesses a patient's abilities and limitations with respect to everyday physical activities. Respondents report limitations on a 5-point scale: 5=Not at all, ..., 3=Somewhat, ..., 1=Cannot do, and abilities to perform activities on a 5-point scale: 5=Without any difficulty, ..., 3=With some difficulty, ..., 1=Unable to do. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 13.5 to 61.9. Higher T-scores represent better outcomes.
Time Frame: At baseline; at week 11 (post-intervention); at week 16 (1 month post intervention)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | LARKSPUR Intervention | Attention Control Condition
Number analyzed (Participants) | 43 | 43
T-score
  Baseline | 36.72 [34.92 to 38.53] | 36.99 [35.28 to 38.69]
  Week 11 (Post-Intervention) | 38.71 [37.39 to 40.04] | 38.46 [37.14 to 39.79]
  Week 16 (1 Month Post-Intervention): number analyzed (Participants) | 41 | 43
  Week 16 (1 Month Post-Intervention) | 39.39 [38.05 to 40.73] | 38.18 [36.86 to 39.51]
Statistical Analysis 1: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 11 (Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PROMIS Physical Functioning scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.792, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-1.63 to 2.13], Standard Error of Mean 0.95 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 2: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PROMIS Physical Functioning scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.209, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = 1.20, 95% CI 2-sided [-0.69 to 3.09], Standard Error of Mean 0.95 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 3: Comparison: LARKSPUR Intervention vs Attention Control Condition; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.151, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = 0.95, 95% CI 2-sided [-0.35 to 2.26], Standard Error of Mean 0.66 — [estimate comment as in outcome 5, analysis 3]

8. Secondary Outcome: Change in Physical Functioning as Measured by PROMIS Fatigue - Short Form 6a (Aim 2)
Description: Fatigue T-scores measured by PROMIS Fatigue Short Form 6a. This 6-item instrument assesses a patient's a patient's level of fatigue over a 7-day recall period. Respondents report fatigue on a 5-point scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 33.4 to 76.8. Lower T-scores represent better outcomes.
Time Frame: At baseline; at week 11 (post-intervention); at week 16 (1 month post intervention)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | LARKSPUR Intervention | Attention Control Condition
Number analyzed (Participants) | 43 | 43
T-score
  Baseline | 66.88 [65.02 to 68.73] | 62.79 [60.68 to 64.89]
  Week 11 (Post-Intervention) | 62.32 [60.25 to 64.40] | 61.55 [59.50 to 63.60]
  Week 16 (1 Month Post-Intervention): number analyzed (Participants) | 41 | 43
  Week 16 (1 Month Post-Intervention) | 61.96 [59.85 to 64.08] | 63.62 [61.57 to 65.67]
Statistical Analysis 1: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 11 (Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PROMIS Fatigue scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.601, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [-2.14 to 3.69], Standard Error of Mean 1.47 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 2: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PROMIS Fatigue scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.269, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = -1.65, 95% CI 2-sided [-4.60 to 1.29], Standard Error of Mean 1.49 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 3: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) in change from Week 11 (Post-Intervention) to Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PROMIS Fatigue scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.116, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = -2.43, 95% CI 2-sided [-5.47 to 0.61], Standard Error of Mean 1.53 — [estimate comment as in outcome 5, analysis 3]

9. Secondary Outcome: Change in Depressive Symptoms as Measured by the Center for Epidemiologic Studies Depression Scale Revised (CESD-R-10) (Aim 2)
Description: The 10-item version of the Center for Epidemiological Studies Depression Scale (CES-D) asks for participants to rate how often over the past week they experienced symptoms associated with depression on a 4-point scale: 0=Rarely or None of the time, 1=Some or Little of the time, 2=Moderately or Much of the time, 3=Most or Almost all the time. CESD-R-10 mean scores range from 0 (rare depressive symptoms) to 4 (depressive symptoms most or almost all the time).
Time Frame: At baseline; at week 11 (post-intervention); at week 16 (1 month post intervention)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LARKSPUR Intervention | Attention Control Condition
Number analyzed (Participants) | 43 | 43
units on a scale
  Baseline | 1.26 [1.09 to 1.43] | 1.19 [1.02 to 1.36]
  Week 11 (Post-Intervention) | 1.13 [1.02 to 1.25] | 1.07 [0.96 to 1.19]
  Week 16 (1 Month Post-Intervention): number analyzed (Participants) | 41 | 43
  Week 16 (1 Month Post-Intervention) | 1.39 [1.27 to 1.51] | 1.26 [1.15 to 1.38]
Statistical Analysis 1: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 11 (Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline CESD-R-10 scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.479, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.10 to 0.22], Standard Error of Mean 0.08 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 2: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline CESD-R-10 scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.126, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.04 to 0.29], Standard Error of Mean 0.08 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 3: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) in change from Week 11 (Post-Intervention) to Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline CESD-R-10 scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.457, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.12 to 0.25], Standard Error of Mean 0.09 — [estimate comment as in outcome 5, analysis 3]

10. Secondary Outcome: Change in Positive Affect as Measured by the Modified Differential Emotions Scale (mDES) (Aim 2)
Description: The modified Differential Emotions Scale (mDES) is a 20-item instrument that measures the extent to which a patient has experienced positive and negative emotions over a chosen time frame; in the version used in this study, we ask for emotions over the past 7 days. Respondents are asked to report the greatest amount of a given emotion on a five-point scale: 0=Not at all, 1=A little bit, 2=Moderately, 3=Quite a bit, 4=Extremely. mDES mean scores range from 0 (not at all experienced positive emotion) to 4 (extremely positive emotion).
Time Frame: At baseline; at week 11 (post-intervention); at week 16 (1 month post intervention)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LARKSPUR Intervention | Attention Control Condition
Number analyzed (Participants) | 43 | 43
units on a scale
  Baseline | 1.94 [1.72 to 2.16] | 1.99 [1.79 to 2.19]
  Week 11 (Post-Intervention) | 2.26 [2.08 to 2.45] | 2.15 [1.96 to 2.34]
  Week 16 (1 Month Post-Intervention): number analyzed (Participants) | 41 | 43
  Week 16 (1 Month Post-Intervention) | 2.49 [2.30 to 2.68] | 2.39 [2.12 to 2.48]
Statistical Analysis 1: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 11 (Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline mDES scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.389, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.15 to 0.38], Standard Error of Mean 0.13 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 2: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline mDES scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.157, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.07 to 0.46], Standard Error of Mean 0.13 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 3: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) in change from Week 11 (Post-Intervention) to Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline mDES scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.593, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.21 to 0.36], Standard Error of Mean 0.14 — [estimate comment as in outcome 5, analysis 3]

11. Secondary Outcome: Change in Positive Affect as Measured by the Positive and Negative Affect Scale (PANAS-GEN) (Aim 2)
Description: The 20-item self-report Positive and Negative Affect Scale (PANAS-GEN) asks participants to describe to what extent they feel different feelings and emotions on average. Respondents answer on a five-point scale: 0=Very slightly or not at all, 1=A little, 2=Moderately, 3=Quite a bit, 4=Extremely. PANAS-GEN mean scores range from 0 (very slightly or not at all positive affect) to 4 (extremely positive affect).
Time Frame: At baseline; at week 11 (post-intervention); at week 16 (1 month post intervention)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LARKSPUR Intervention | Attention Control Condition
Number analyzed (Participants) | 43 | 43
units on a scale
  Baseline | 1.94 [1.72 to 2.16] | 1.99 [1.79 to 2.19]
  Week 11 (Post-Intervention) | 1.88 [1.71 to 2.06] | 1.90 [1.72 to 2.07]
  Week 16 (1 Month Post-Intervention): number analyzed (Participants) | 41 | 43
  Week 16 (1 Month Post-Intervention) | 2.04 [1.86 to 2.22] | 1.98 [1.80 to 2.16]
Statistical Analysis 1: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 11 (Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PANAS-GEN scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.933, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.26 to 0.24], Standard Error of Mean 0.13 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 2: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PANAS-GEN scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.642, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.19 to 0.31], Standard Error of Mean 0.13 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 3: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) in change from Week 11 (Post-Intervention) to Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PANAS-GEN scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.577, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.18 to 0.32], Standard Error of Mean 0.12 — [estimate comment as in outcome 5, analysis 3]

12. Secondary Outcome: Change in Stress Appraisal as Measured by the Perceived Stress Scale (Aim 2)
Description: The 10-item version of the Perceived Stress Scale (PSS) assesses the perception of stress over the previous month. Respondents report how often they have experienced perceived stress on a five-point scale: 0=Never, 1=Almost never, 2=Sometimes, 3=Fairly often, 4=Very often. PSS mean scores range from 0 (experienced no or minimal stress) to 4 (experienced very frequent stress).
Time Frame: At baseline; at week 11 (post-intervention); at week 16 (1 month post intervention)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LARKSPUR Intervention | Attention Control Condition
Number analyzed (Participants) | 43 | 43
units on a scale
  Baseline | 1.87 [1.65 to 2.09] | 1.65 [1.46 to 1.83]
  Week 11 (Post-Intervention) | 1.55 [1.40 to 1.71] | 1.65 [1.49 to 1.81]
  Week 16 (1 Month Post-Intervention): number analyzed (Participants) | 41 | 43
  Week 16 (1 Month Post-Intervention) | 1.48 [1.32 to 1.64] | 1.69 [1.54 to 1.85]
Statistical Analysis 1: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 11 (Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PSS scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.403, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.32 to 0.13], Standard Error of Mean 0.11 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 2: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) at Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PROMIS PSS scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.062, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.44 to 0.01], Standard Error of Mean 0.11 — The estimated Mean Difference compares the LARKSPUR intervention minus the Attention Control
Statistical Analysis 3: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) in change from Week 11 (Post-Intervention) to Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and two time points (Week 11, Week 16) and their interaction adjusting for baseline PSS scores. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.269, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.33 to 0.09], Standard Error of Mean 0.11 — [estimate comment as in outcome 5, analysis 3]

13. Other Pre Specified Outcome: Change in Affective Reactivity to Stress as Measured by the Daily Modified Differential Emotions Scale (mDES)
Description: Positive affective reactivity measured by the modified Differential Emotions Scale (mDES). Upon completion of each study assessment, participants completed the mDES daily for one week, for a total of three 7-day-long periods. The mDES is a 20-item instrument that measures the extent to which a patient has experienced positive (10 items) and negative (10 items) emotions over a chosen time frame; in the version used in this survey, we ask for emotions over the past 24 hours. Respondents are asked to report the greatest amount of positive affect on a five-point scale: 0=Not at all, 1=A little bit, 2=Moderately, 3=Quite a bit, 4=Extremely. mDES mean scores were computed over the 10 items, ranging from 0 (not at all positive) to 4 (extremely positive).
Time Frame: At baseline, at week 11 (post-intervention); at week 16 (1 month post intervention)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LARKSPUR Intervention | Attention Control Condition
Number analyzed (Participants) | 43 | 43
units on a scale
  Baseline | 1.68 [1.47 to 1.87] | 1.70 [1.50 to 1.90]
  Week 11 (Post-Intervention) | 1.83 [1.62 to 2.03] | 1.66 [1.46 to 1.86]
  Week 16 (1 Month Post-Intervention): number analyzed (Participants) | 41 | 43
  Week 16 (1 Month Post-Intervention) | 1.79 [1.59 to 1.99] | 1.64 [1.44 to 1.84]
Statistical Analysis 1: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) in change from Baseline to Week 11 (Post-Intervention) was tested using a mixed effects model with two treatment groups and three time points (Baseline, Week 11, Week 16) and their interaction while accounting for heterogeneous (random slopes) linear daily trends. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.003, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = 0.20, 95% CI 2-sided [0.07 to 0.33], Standard Error of Mean 0.07 — The estimated Mean Difference (Net) compares the change for the LARKSPUR intervention (Week 11 minus Baseline) minus the change for the Attention Control (Week 11 minus Baseline)
Statistical Analysis 2: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) in change from Baseline to Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and three time points (Baseline, Week 11, Week 16) and their interaction while accounting for heterogeneous (random slopes) linear daily trends. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.006, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = 0.18, 95% CI 2-sided [0.05 to 0.31], Standard Error of Mean 0.07 — The estimated Mean Difference (Net) compares the change for the LARKSPUR intervention (Week 16 minus Baseline) minus the change for the Attention Control (Week 16 minus Baseline)
Statistical Analysis 3: Comparison: LARKSPUR Intervention vs Attention Control Condition; The treatment difference (LARKSPUR Intervention vs. Attention Control) in change from Week 11 (Post-Intervention) to Week 16 (1 Month Post-Intervention) was tested using a mixed effects model with two treatment groups and three time points (Baseline, Week 11, Week 16) and their interaction while accounting for heterogeneous (random slopes) linear daily trends. Sample size was chosen based on feasibility indicators (recruitment, retention, adherence) rather than on formal power analyses; Test type: Superiority; p = 0.796, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.15 to 0.12], Standard Error of Mean 0.07 — [estimate comment as in outcome 5, analysis 3]

14. Other Pre Specified Outcome: Change in Affective Reactivity to Stress as Measured by the Daily Inventory of Stressful Events (DISE)
Description: Affective reactivity to stress measured by the Daily Inventory of Stressful Events (DISE). Upon completion of each study assessment, patients completed the DISE daily for one week, for a total of three 7-day-long periods. The DISE is a 7-item self-report instrument in which participants report whether stressful events (argument, work or school stress, home stress, discrimination, close friend stress, other stressors) have occurred within the past 24 hours, indicating "yes" or "no" accordingly for each item. Item scores are averaged, ranging from 0=no stress to 1=highest stress. Higher scores indicate worse outcomes.
Time Frame: At baseline, at week 11 (post-intervention); at week 16 (1 month post intervention)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LARKSPUR Intervention | Attention Control Condition
Number analyzed (Participants) | 43 | 43
units on a scale
  Baseline | 0.21 [0.16 to 0.26] | 0.17 [0.12 to 0.22]
  Week 11 (Post-Intervention) | 0.21 [0.16 to 0.26] | 0.17 [0.12 to 0.21]
  Week 16 (1 Month Post-Intervention): number analyzed (Participants) | 41 | 43
  Week 16 (1 Month Post-Intervention) | 0.19 [0.14 to 0.24] | 0.16 [0.11 to 0.20]
Statistical Analysis 1: Comparison: LARKSPUR Intervention vs Attention Control Condition; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.758, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.03 to 0.05], Standard Error of Mean 0.02 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: LARKSPUR Intervention vs Attention Control Condition; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = 0.880, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.04 to 0.04], Standard Error of Mean 0.02 — [estimate comment as in outcome 13, analysis 2]
Statistical Analysis 3: Comparison: LARKSPUR Intervention vs Attention Control Condition; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p = 0.652, Mixed Models Analysis — The threshold for statistical significance was 0.05; Degrees of freedom and standard error estimates were adjusted using the Kenward-Roger (1997) method; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.05 to 0.03], Standard Error of Mean 0.02 — [estimate comment as in outcome 5, analysis 3]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 4 months per participant.
Description: This was an on-line behavioral intervention with assessments also done remotely. The study was deemed minimal risk to participants.
Arm/Group | LARKSPUR Intervention | Attention Control Condition
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/46
Other Adverse Events (participants affected / at risk) | 0/49 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT04869345/Prot_001.pdf
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT04869345/SAP_002.pdf
  • Informed Consent Form (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT04869345/ICF_003.pdf